CLINICAL TRIAL: NCT04054687
Title: Intranasal TXA for Anterior Epistaxis in the Emergency Department
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to coronavirus pandemic
Sponsor: Mercy Health Ohio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 19-001
Record Dates: First submitted 2019-03-12; First posted 2019-08-13 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Epistaxis
MeSH Terms: conditions — Epistaxis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TXA (Experimental): Research participants in the experimental group will receive one dose of 100mg/mL TXA soaked in a cotton pledget in the bleeding nare for a total of 15 minutes.
  Interventions: Drug: Tranexamic Acid
- Saline (Placebo Comparator): Research participants in the placebo group will receive one dose of normal saline (0.9%) soaked in a cotton pledget in the bleeding nare for a total of 15 minutes.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Enrolled patients will be placed in one of two groups: either the group receiving a cotton pledget soaked in (0.9%) saline or (100mg/1mL) TXA. Patients will initially be asked to gently blow their nose to remove any clots. Group 1 will receive the saline soaked pledget. After fifteen minutes the pledget will be removed. If patient continues to bleed within a reevaluation period of fifteen minutes, this will be deemed a 'failure' and the examiner will pack the nose with the method of his or her choice. Group 2 will receive the TXA soaked pledget and the procedure will continue like Group 1.
  Other Names: TXA
  Arms: TXA
Other: Placebo — This group will receive pledget soaked in saline. Protocol will continue as with TXA group.
  Other Names: Normal saline
  Arms: Saline

SUMMARY:
The objective of this study is to evaluate the efficacy of and patient satisfaction with the use of intranasal tranexamic acid (TXA) for anterior nosebleeds in the emergency department (ED).

DETAILED DESCRIPTION:
Pledget soaked in either saline or TXA will be applied to the bleeding nare of the patient presenting with anterior epistaxis. After fifteen minutes, the pledget will be removed and patient reassessed.

Informed consent will be obtained prior to patient enrollment.

Enrolled patients will be placed in one of two groups: either the group receiving a cotton pledget soaked in (0.9%) saline or (100mg/1mL) TXA. Patients will initially be asked to gently blow their nose to remove any clots. Group 1 will receive the saline soaked pledget. After fifteen minutes the pledget will be removed. If patient continues to bleed within a reevaluation period of fifteen minutes, this will be deemed a 'failure' and the examiner will pack the nose with the method of his or her choice. Group 2 will receive the TXA soaked pledget and the procedure will continue like Group 1.

Patient satisfaction will be assessed in both groups during ED stay and one week after ED stay.

ELIGIBILITY:
Inclusion criteria:

• Patients 18 years and older with anterior epistaxis

Exclusion criteria:

* Patients with inability to give consent
* Patients without a working telephone number
* Patients lacking the mental capacity to make their own decisions
* Patients with posterior epistaxis
* Epistaxis following major trauma
* Patients with known bleeding disorder like hemophilia and thrombocytopenia
* Prisoners
* Patients hemodynamically unstable
* Pregnant patients
* Patients with a known allergy to TXA
* Patients with a visibly bleeding vessel
* Those recently post-op nasal/sinus surgery (within ten days) will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Bleeding cessation | 15 minutes
  After 15 minutes of patient receiving either pledget filled TXA or placebo, bleeding will be assessed

SECONDARY OUTCOMES:
Patient satisfaction: 10 point scale | Before ED discharge (up to 24 hours) and 1 week after ED discharge
  Patient satisfaction will be assessed at the end of the emergency department encounter, and then again via telephone call one week after discharge using a 10 point scale
Bleeding cessation | 1 week
  Patients will be contacted 1 week after ED discharge to determine whether there was a recurrence of his/her epistaxis

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Barreiro, Study Chair — Mercy Health
Locations (2):
- United States (2):
  - St Elizabeth Boardman Hospital, Boardman, Ohio
  - St Elizabeth Youngstown, Youngstown, Ohio

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT04054687/Prot_SAP_000.pdf